CLINICAL TRIAL: NCT06337071
Title: A Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of the ACYW135 Meningococcal Polysaccharide Conjugate Vaccine in People Aged 3 Months to 15 Years Old in a Randomized, Double-blind, Parallel Controlled Design
Brief Title: A Study of the ACYW135 Meningococcal Polysaccharide Conjugate Vaccine
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aimei Vacin BioPharm (Zhejiang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AM2023MCV4Ⅱ
Record Dates: First submitted 2024-03-13; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Meningococcal Meningitis
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Experimental Group 2~15 years (Experimental): 2~15 years old participants who vaccinated by experimental vaccine
  Interventions: Biological: ACYW135 Meningococcal Polysaccharide Conjugate Vaccine
- Control Group 2~15 years (Active Comparator): 2~15 years old participants who vaccinated by control vaccine 2
  Interventions: Biological: ACYW135 Meningococcal Polysaccharide Vaccine
- Experimental Group 6~23 months(0,1) (Experimental): 6~23 months old participants who vaccinated by experimental vaccine at month 0 and 1
  Interventions: Biological: ACYW135 Meningococcal Polysaccharide Conjugate Vaccine
- Control Group 6~23 months(0,1) (Active Comparator): 6~23 months old participants who vaccinated by control vaccine 1 at month 0 and 1
  Interventions: Biological: ACYW135 Meningococcal Polysaccharide Conjugate Vaccine
- Experimental Group 6~23 months(0,3) (Experimental): 6~23 months old participants who vaccinated by experimental vaccine at month 0 and 3
  Interventions: Biological: ACYW135 Meningococcal Polysaccharide Conjugate Vaccine
- Control Group 6~23 months(0,3) (Active Comparator): 6~23 months old participants who vaccinated by control vaccine 1 at month 0 and 3
  Interventions: Biological: ACYW135 Meningococcal Polysaccharide Conjugate Vaccine
- Experimental Group 3~5 months (Experimental): 3~5 months old participants who vaccinated by experimental vaccine at month 0, 1, 2 for primary vaccination, and vaccinated by experimental vaccine at 12-month old for booster vaccination
  Interventions: Biological: ACYW135 Meningococcal Polysaccharide Conjugate Vaccine
- Control Group 3~5 months (Active Comparator): 3~5 months old participants who vaccinated by control vaccine 1 at month 0, 1, 2 for primary vaccination, and vaccinated by control vaccine at 12-month old for booster vaccination
  Interventions: Biological: ACYW135 Meningococcal Polysaccharide Conjugate Vaccine

INTERVENTIONS:
Biological: ACYW135 Meningococcal Polysaccharide Conjugate Vaccine — ACYW135 Meningococcal Polysaccharide Conjugate Vaccine was produced by meningococcal polysaccharide from group A, C, Y, W135 and conjugated protein CRM197.
  Arms: Control Group 3~5 months; Control Group 6~23 months(0,1); Control Group 6~23 months(0,3); Experimental Group 2~15 years; Experimental Group 3~5 months; Experimental Group 6~23 months(0,1); Experimental Group 6~23 months(0,3)
Biological: ACYW135 Meningococcal Polysaccharide Vaccine — ACYW135 Meningococcal Polysaccharide Vaccine was produced by meningococcal polysaccharide from group A, C, Y, W135.
  Arms: Control Group 2~15 years

SUMMARY:
The purpose of this study was to explore the safety and immunogenicity of the experimental vaccine compared with the control vaccines. It is planed to enroll a total of 1,200 subjects, including 300 subjects in each of the 3-5 months old, 6-11 months old, 12-23 months old and 2-15 years old groups, who will be randomly assigned to the trial in a 1:1 ratio to study group or control group. The 3-5 month-old group will have three doses vaccination at 0, 1 and 2 month, and a booster dose at 12 months of age; the 6-11month-old and 12-23 month-old groups will each have total two doses vaccination; the 2-15 year-old group will have one dose vaccination.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the safety and immunogenicity of the experimental vaccine(ACYW135 Meningococcal Polysaccharide Conjugate Vaccine) compared with the control vaccines(ACYW135 Meningococcal Polysaccharide Conjugate Vaccine and ACYW135 Meningococcal Polysaccharide Vaccine). It is planed to enroll a total of 1,200 subjects, including 300 subjects in each of the 3-5 months old, 6-11 months old, 12-23 months old and 2-15 years old groups, who will be randomly assigned to the trial in a 1:1 ratio to study group or control group. The 3-5 month-old group will have three doses vaccination at 0, 1 and 2 month, and a booster dose at 12 months of age; the 6-11month-old and 12-23 month-old groups will each have total two doses vaccination(at month 0, 1 or at month 0, 3); the 2-15 year-old group will have one dose vaccination. The immunogenicity and immune persistence will be evaluated by rabbit complement serum bactericidal assay.

ELIGIBILITY:
Inclusion Criteria:

* 3~5 months old:

  1. 3~5 months old;
  2. The subject's legal guardian voluntarily agrees to his or her child's participation in this trial and signs an informed consent form;
  3. The subject and/or the subject's legal guardian can comply with the relevant requirements of the clinical trial protocol;
  4. Have not vaccinated by any meningococcal vaccine in the past.
* 6~23 months old:

  1. 6~23 months old;
  2. The subject's legal guardian voluntarily agrees to his or her child's participation in this trial and signs an informed consent form;
  3. The subject and/or the subject's legal guardian can comply with the relevant requirements of the clinical trial protocol;
  4. Have not vaccinated by any other meningococcal vaccines except meningococcal group A polysaccharide vaccine in the past. If have 1 dose vaccinated of meningococcal group A polysaccharide vaccine, it will be 3 months or more separated from the previous dose of meningococcal group A polysaccharide vaccine. If two doses of meningococcal group A polysaccharide vaccine have been vaccinated, the interval between the last dose of meningococcal group A polysaccharide vaccine should be more than 6 months or more.
* 2~15 years old:

  1. 2~15 years old;
  2. The subject's legal guardian voluntarily agrees to his or her child's participation in this trial and signs an informed consent form (subjects aged 8-15 years old are also required to sign an informed consent form);
  3. The subject and/or the subject's legal guardian can comply with the relevant requirements of the clinical trial protocol; Subjects aged 2 to 6 years old have not previously been vaccinated with any meningococcal vaccine other than meningococcal polysaccharide vaccine, and the interval between the previous dose of meningococcal polysaccharide vaccine and vaccination should be more than 12 months or more; 7~15 years old participants have not received any meningococcal vaccine in the past 3 years.

Exclusion Criteria:

1. The temperature before vaccination on the day of vaccination is >37.0℃;
2. Have a history of invasive disease caused by meningococci confirmed by culture;
3. Have a history of severe allergic reactions that require medical intervention (such as oral and throat swelling, dyspnea, hypotension or shock caused by allergies); have a history of allergies to vaccines or vaccine components (especially those allergic to diphtheria toxoid), and have concerns about vaccination History of other serious adverse reactions;
4. Those with a clearly diagnosed history of thrombocytopenia or other coagulation disorders, which may cause contraindications for intramuscular injection;
5. Suffer from acute disease or acute attack of chronic disease within 3 days before vaccination;
6. Have a history of epilepsy, progressive neurological disease, Guillain-Barré syndrome, convulsions (except simple febrile convulsions) and mental illness;
7. Known or suspected immunological dysfunction, including immunosuppressant treatment (radiation therapy, chemotherapy, corticosteroids, antimetabolites, cytotoxic drugs), human immunodeficiency virus (HIV) infection, etc.;
8. Known severe congenital malformations; suffering from developmental disabilities or clinically diagnosed serious chronic diseases (such as Down syndrome, diabetes, sickle cell anemia or neurological diseases);
9. Known or suspected to have serious diseases that are judged by the researcher to affect vaccination, including respiratory diseases, digestive system diseases, endocrine system diseases, immune system diseases, cardiovascular diseases, liver and kidney diseases, malignant tumors, skin diseases, etc. ;
10. Long-term use (continuous use for ≥14 days) of immunosuppressants or other immunomodulatory drugs (such as corticosteroids: prednisone or similar drugs) within 6 months before vaccination with the experimental vaccine, but local use (such as ointments, eye drops, inhalants, or nasal sprays), topical administration should not exceed the dosage recommended in the label;
11. Have received blood products including gamma globulin or immune globulin treatment within 3 months before vaccination (<3 months);
12. Asplenia or functional asplenia, asplenia or splenectomy caused by any condition;
13. Have been vaccinated with live attenuated vaccines within 14 days (including 14 days) before vaccination, and have been vaccinated with other subunits, inactivated vaccines or recombinant protein vaccines other than live attenuated vaccines within 7 days (including 7 days);
14. Currently participating in or planning to participate in other drug clinical trials during the entire trial period after receiving the experimental vaccine;
15. Any situation that the researcher believes may affect the evaluation of the trial.

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity 1 | 30 days after primary vaccination
  To evaluate the positive conversion rate and geometric mean titer (GMT) of meningococcal serum bactericidal activity (rSBA) antibodies for meningococcal groups A, C, Y, and W135 at 30 days in 3~5 months old participants after primary vaccination
Immunogenicity 2 | 30 days after two doses vaccination
  To evaluate the positive conversion rate and geometric mean titer (GMT) of meningococcal serum bactericidal activity (rSBA) antibodies for meningococcal groups A, C, Y, and W135 at 30 days in 6~23 months old participants after two doses vaccination
Immunogenicity 3 | 30 days after one dose vaccination
  To evaluate the positive conversion rate and geometric mean titer (GMT) of meningococcal serum bactericidal activity (rSBA) antibodies for meningococcal groups A, C, Y, and W135 at 30 days in 2~15 years old participants after one dose vaccination
Safety 1 | 30 days after each dose vaccination
  The incidence of adverse events (AEs)/vaccination-related AEs on days 0 to 30 after each dose of immunization for subjects in each age group

SECONDARY OUTCOMES:
Immunogenicity 4 | 30 days after booster vaccination
  To evaluate the positive rate of serum bactericidal activity (rSBA) antibodies against meningococcal groups A, C, Y and W135 (ratio of antibody titers ≥1:8), ratio of antibody titer ≥1:128, geometric mean growth factor (GMFI) in 3~5 months old participants after primary vaccination
Immunogenicity 5 | Before booster vaccination
  To evaluate the serum bactericidal activity (rSBA) antibody GMT, positivity rate and rate of antibody titer ≥1:128 subjects in 3~5 months old participants before booster vaccination
Immunogenicity 6 | 30 days after booster vaccination
  To evaluate the serum bactericidal activity (rSBA) antibody positive conversion rate, GMT, GMFI, positivity rate, and rate of antibody titer≥ 1:128 ratio in 3~5 months old participants after booster vaccination
Immunogenicity 7 | 30 days after booster vaccination
  To evaluate the positive rate of serum bactericidal activity (rSBA) antibodies against meningococcal groups A, C, Y and W135 (ratio of antibody titers ≥1:8), ratio of antibody titer ≥1:128, geometric mean growth factor (GMFI) in 6~23 months old participants after two doses vaccination
Immunogenicity 8 | 30 days after vaccination
  To evaluate the positive rate of serum bactericidal activity (rSBA) antibodies against meningococcal groups A, C, Y and W135 (ratio of antibody titers ≥1:8) and ratio of antibody titer ≥1:128 in 6~23 months old participants after vaccination
Immune persistence 1 | 6 months after booster vaccination
  To evaluate the serum bactericidal activity (rSBA) antibody positivity rate, rate of antibody titer ≥1:128 and GMT in 3~5 months old participants after booster vaccination
Immune persistence 2 | 6 months, 12 months
  To evaluate the serum bactericidal activity (rSBA) antibody positivity rate, rate of antibody titer ≥1:128 and GMT in 6~23 months old participants after two doses vaccination
Safety 2 | 30 days after each dose vaccination
  AEs/vaccination-related AEs are divided into doses, severity, vaccination site and non-vaccination site, and system organs (SOC) classification and incidence of each preferred term (PT) symptom after each dose vaccination
Safety 3 | 6 months after primary vaccination and 30 days after booster vaccination
  The occurrence of serious adverse events (SAE) in each group of subjects aged 3 to 5 months from the first dose vaccination to 6 months after primary vaccination and within 30 days after booster vaccination
Safety 4 | 6 months after all doses vaccination
  The occurrence of serious adverse events (SAE) in each group of subjects aged 2~15 years and 6~23 months from the first dose vaccination to 6 months after all doses vaccination

CONTACTS AND LOCATIONS:
Overall Officials: ZHENG Yan, Principal Investigator — YUNNAN CENTER FOR DISEASE CONROL AND PREVENTION
Locations (1):
- Yunnan Center For Disease Control and Prevention, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No